CLINICAL TRIAL: NCT01668810
Title: The Third Survey on China Psychotropic Prescription for Schizophrenia, Depression and Bipolar Disorder
Brief Title: The Third Survey of Prescription Pattern of Psychotropic Drugs in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Principal Investigator, Si Tianmei, Professor, Peking University
Other Study IDs: RISSCH4255
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-07

CONDITIONS: Prescription
Keywords: prescription; schizophrenia; depression; bipolar disorder
MeSH Terms: conditions — Schizophrenia; Depression; Bipolar Disorder

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (10):
- Beijing region: include six hospitals
- Guangdong Province: include 3 hospitals
- Jiangsu province: include 3 hospitals
- Hebei province: include 6 hospitals
- Hubei Province: include 7 hospitals
- Shanxi province: include 3 hospitals
- Jiangxi province: include 3 hospitals
- Jilin province: include 6 hospitals
- Sichuan province: include 3 hospitals
- Shaanxi province: include 3 hospitals

SUMMARY:
The investigators aimed to examine the psychotropic prescription pattern in China.

ELIGIBILITY:
Inclusion Criteria: aged 18-65, inpatient or outpatient, Patient must be willing and able to give written informed consent,the patient suffers from schizophrenia or depression or bipolar disorder -

Exclusion Criteria:aged<18or aged>65

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: schizophrenia, depression and bipolar disorder patients
Sampling Method: Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-09 (Estimated); Study Completion 2013-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Xin Yu, MD., Study Chair — Peking University
Locations (1):
- Institute of mental health, Peking University, Beijing, Beijing Municipality, China